CLINICAL TRIAL: NCT04893785
Title: A Phase II Single Arm Interventional Trial Evaluating the Activity and Safety of Combination Between Cabozantinib and Temozolomide in Lung and GEP-NENS Progressive After Everolimus, Sunitinib or PRRT (CABOTEM)
Brief Title: A Trial Evaluating the Activity and Safety of Combination Between Cabozantinib and Temozolomide in Lung and GEP-NENS Progressive After Everolimus, Sunitinib or PRRT (CABOTEM)
Acronym: CABOTEM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CABOTEM
Record Dates: First submitted 2021-05-14; First posted 2021-05-20 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Lung Neuroendocrine Neoplasm; GEP Neuroendocrine Tumor
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor | interventions — cabozantinib; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cabozantinib and Temozolomide (Experimental): All patients will receive:
  * Cabozantinib 40 mg os QD
  * Temozolomide 100 mg/m2/day seven days followed by seven days of stop (regimen one week on / one week off).
  Interventions: Drug: Cabozantinib and Temozolomide

INTERVENTIONS:
Drug: Cabozantinib and Temozolomide — Patients enrolled will receive study medication until disease progression, unacceptable toxicity, withdrawal of consent or death, whichever comes first.
  Patients will be required to attend clinic on Day 1, Day 8, Day 14 and Day 22 of every 4 week cycle.
  Patients will return to clinic at 30 days (+/- 5 days) of their last dose of cabozantinib or temozolomide (whichever is discontinued last), for an end of treatment visit.
  Following their end of treatment visit patients will be followed-up 3-monthly during routine clinic appointments to collect data on further anti-cancer treatment and survival. Follow-up will continue until 6 months after the last patient stops study treatment or up to 18 months after the last patient is randomised, whichever is sooner.

SUMMARY:
The aim of CABOTEM study is to demonstrate the safety and activity of the Cabozantinib and Temozolomide combination in Lung and GEP-NENs patients, progressing after a first line therapy, including target therapies (everolimus, sunitinib) and / or chemotherapy, in the approved setting.

DETAILED DESCRIPTION:
Neuroendocrine neoplasms (NENs) are a heterogeneous group of neoplasms, mainly originating from the gastro-entero-pancreatic system and the lung. Molecular targeted therapy of NENs with the mTOR inhibitor everolimus is currently approved for GEP-Lung NENs and with the multi-tyrosine kinase inhibitor (multiTKI) sunitinib (VEGFR, PDGFR, KIT) for PAN-NENs. There is still an unmet need for further medical therapies including novel targeted therapies, the knowledge of the data on the role of the sequences of the therapies and the definition of new biological predictors of outcome and prognosis.

Cabozantinib targets VEGF receptors, MET, AXL, and RET. Cabozantinib is an oral, potent inhibitor of mesenchymal-epithelial transition factor (MET), VEGF receptor 2 (VEGFR2), and RET that produces robust antiangiogenic, antiproliferative, and antiinvasive effects in preclinical models. It has been shown to improve outcomes in advanced renal cell carcinoma patients in both the first-line and second-line settings and is also approved for progressive, metastatic medullary thyroid cancer.

Recent studies have suggested that activation of the MET signalling pathway may also play a role in the growth of neuroendocrine tumours. Increased expression of MET correlates with decreased overall survival in pancreatic neuroendocrine tumours. In preclinical pancreatic neuroendocrine tumour models, various multi-TKIs with combined anti-VEGF and anti-MET efficacy have shown enhanced angiogenesis inhibition, as well as suppression of tumour invasion and metastasis . Given the strong theoretical rationale for combining anti-VEGF and anti-MET activity in neuroendocrine tumours, in USA will start randomized, double-blinded phase III trial, named CABINET to evaluate the effects in terms of PFS in patients with advanced neuroendocrine tumours after progression on everolimus.

In an on-going clinical trial, Chan et al. showed, in patients with progressive, well differentiated, grade 1-2 carcinoid and treated with cabozantinib 60 mg po qd and without limit to prior therapy, 21.8 mo (95% CI, 8.5-32.0 mo) of mPFS in pts with pNET and 31.4 mo (95% CI, 8.5 mo-NR) in pts with carcinoid . In this study pNET achieved PR (ORR 15%, 95% CI 5-36%); 15/20 had SD. 6/41 pts with carcinoid achieved PR (ORR 15%, 95% CI 7-28%); 26/41 had SD.

The front-line treatment of advanced NENs depends on many clinical and pathological factors but there are no standard second-line therapies when the disease progress. Although data for temozolomide (TMZ)-based chemotherapy are still evolving, this treatment may replace STZ-based regimens in PAN-NENs due to its better tolerability and side effect profile. In addition, there is evidence that TMZ could also be used in the subgroup of well-differentiated G3 NETs. There is less clear-cut evidence of a benefit for chemotherapy in intestinal NETs, but still evolving data suggest that TMZ may be efficacious in particular patients. In our experiences, an intermittent schedule of metronomic TMZ is effective and safe in patients with advanced progressive G2-G3 NEN, showing to be a feasible second line treatment in this setting. This schedule has been also investigated by Chan et al. in 34 patients with advanced neuroendocrine tumors demonstrating a good safety profile. D.Shiff et al. demonstrated that cabozantinib at a dose of 40/60 mg daily plus TMZ for patients with newly diagnosed high-grade glioma was generally well tolerated even with the addition of radiotherapy, and also demonstrated no pharmacokinetic interactions with concurrent TMZ. Both mRNA and protein levels of c-Met were significantly associated with tumour grade progression and inversely correlated with overall and progression-free survival in high-grade gliomas. c-Met seems an independent prognostic marker in glioblastoma patients and further analysis in vitro revealed that downregulating the expression of c-Met dramatically inhibited cell migration and invasion capacities, enhanced sensitivity to TMZ chemotherapy . Cabozantinib downregulating c-MET pathway can induce, in addition to antiangiogenic and antiproliferative effects, also an increased sensitivity to Temozolomide.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years and older patients.
2. Signed informed consent prior to initiation of any study-specific procedures or treatment, as confirmation of the patient's awareness and willingness to comply with the study requirements.
3. Documented histological or cytological diagnosis of well differentiated Lung and GEP-NENs (NET G1, NET G2, NET G3 in WHO 2017 classification) progressing after a first line of therapy with SSAs, sunitinib, everolimus, chemotherapy and/or PRRT or documented histological or cytological diagnosis of Large cells neuroendocrine carcinoma patients with Ki67< 55% progressed after platinum-based first line chemotherapy.
4. Subjects must have evidence of progressed disease, radiologically documented in the 12 months previous study entry.
5. Subjects must have evidence of measurable disease as determined by the investigator. Target lesions must have shown evidence of disease progression by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1 criteria in the 12 months prior to study entry. Patients must have measurable disease per RECIST 1.1 by computer tomography (CT) scan or magnetic resonance imaging (MRI). Gallium 68 PET Scan can be considered useful before and during the treatment.
6. Subject must have adequate swallowing capacity.
7. Subjects with functional (associated with a clinical hormone syndrome) and non functional tumors are eligible for the study.
8. The concurrent use of somatostatin analogues is allowed provided that the patient has been on a stable dose for at least two months.
9. At least 4 weeks of wash-out from previous targeted therapies.
10. At least 6 months of wash-out from previous PRRT treatment.
11. Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0-2.
12. Subjects must have adequate organ function, including the following:
13. Bone marrow reserve consistent with: absolute neutrophil count (ANC) ≥1.5 x109/L; platelet count ≥ 100 x 109/L; haemoglobin ≥ 9 g/dL;
14. Hepatic: total bilirubin ≤ 1.5 x upper limit of normal (ULN), transaminases (aspartate aminotransferase/serum glutamic oxaloacetic transaminase [AST/SGOT] and alanine aminotransferase/serum glutamic pyruvic transaminase [ALT/SGPT]) ≤ 2.5 x ULN (< 5 x ULN if liver metastases are present);
15. Renal: normal serum creatinine or calculated creatinine clearance ≥ 60 mL/min (Cockroft-Gault formula);
16. Recovery from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy.
17. Estimated life expectancy of ≥12 weeks
18. Sexually active fertile female subjects must agree to use effective contraceptive methods during the course of the study and for 4 months after the last dose of study treatment. While sexually active fertile male subjects must agree to use effective contraceptive methods during the course of the study and up to 6 months after the last dose of study treatment;
19. For women of child-bearing potential, negative serum pregnancy test within 14 days prior to the first study drug administration;
20. Ability to understand and willingness to sign informed consent form prior to initiation of any study procedures and willingness to comply with the study requirements.

Exclusion Criteria:

1. Receipt of any type of anticancer therapy within 4 weeks before study entry.
2. Previous treatment with Temozolomide or cabozantinib
3. Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before recruitment.
4. Previous PRRT treatment: Systemic treatment with radionuclides within 6 months before study entry.
5. Subjects with clinically relevant ongoing complications from prior radiation therapy and/or surgery are not eligible.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before study entry
7. Concomitant anticoagulation at therapeutic doses with oral anticoagulants or platelet inhibitors.
8. Chronic hepatitis B infection (both active or not).
9. Chronic treatment with corticosteroids or other immuno-suppressive agents.
10. Serious illness other than cancer including, but not limited to, the following conditions:

    1. Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation: i.e. Tumors invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis or acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction ii. Abdominal fistula, GI perforation, bowel obstruction, intra-abdominal abscess within 6 months before recruitment. Note: Complete healing of an intra-abdominal abscess must be confirmed prior to recruitment.
    2. Cavitating pulmonary lesion(s) or endobronchial disease
    3. Lesion invading a major blood vessel including, but not limited to: inferior vena cava, pulmonary artery, or aorta. Subjects with lesions invading the portal vasculature are eligible.
    4. Clinically significant bleeding risk including the following within 3 months of recruitment:

       hematuria, hematemesis, hemoptysis of >0.5 teaspoon (>2.5 mL) of red blood, or other signs indicative of pulmonary hemorrhage, or history of other significant bleeding if not due to reversible external factors
    5. Other clinically significant disorders such as:

    I. Active infection requiring systemic treatment, known infection with human immunodeficiency virus (HIV), or known acquired immunodeficiency syndrome (AIDS)-related illness. II. Serious non-healing wound/ulcer/bone fracture III. Malabsorption syndrome IV. Uncompensated/symptomatic hypothyroidism V. Requirement for hemodialysis or peritoneal dialysis VI. History of solid organ transplantation
11. Uncontrolled congestive heart failure (NYHA II, III, IV). Patients with history of congestive heart failure who do not violate this exclusion criterion will undergo an evaluation of their cardiac ejection fraction prior to recruitment, preferably via gated equilibrium radionuclide ventriculography. The results from an earlier assessment (not exceeding 30 days prior to recruitment) may substitute the evaluation at the discretion of the Investigator, if no clinical worsening is noted. The patient's measured cardiac ejection fraction in these patients must be >40% before recruitment.
12. QTcF > 470 msec for females and QTcF > 450 msec for males or congenital long QT syndrome.
13. Patients with rare hereditary problems of galattose intolerance, congenital lactase deficiency or glucose - galattose malabsorption.
14. Major surgery within 3 months before study entry. Complete wound healing from major surgery must have occurred 1 month before study entry and from minor surgery at least 10 days before study entry.
15. Pregnant or lactating females.
16. History of another malignancy within 2 years before study entry, except for superficial skin cancers.
17. Serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions that could interfere with subject's safety, obtaining informed consent or compliance to the study procedures.
18. Patients on chronic treatment with drugs that are contraindicated to with cabozantinib and temozolomide treatment according to the SmPC of each product.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To assess the efficacy of the combination of cabozantinib and one-week-on/one-week-off temozolomide, based on overall response rate (ORR). | Up to 42 months
  Overall Response Rate (ORR) (as assessed by RECIST v1.1) defined by complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
To assess the activity of the combination of cabozantinib and one-week-on one-week-off temozolomide according to Progression Free Survival (PFS) | Up to 42 months
  PFS (as assessed by RECIST v1.1) defined as time from study entry to first evidence of disease progression or death due to any cause.
To assess the activity of the combination of cabozantinib and one-week-on one-week-off temozolomide according to Clinical Benefit Rate (CBR) | Up to 42 months
  CBR (as assessed by RECIST v1.1) defined by complete response (CR) or partial response (PR) or stable disease (SD).
To assess the activity of the combination of cabozantinib and one-week-on one-week-off temozolomide according to Overall Survival (OS) | Up to 42 months
  OS defined as time from study entry to death due to any cause or to study termination
To assess the activity of the combination of cabozantinib and one-week-on one-week-off temozolomide according to duration of response (DOR) | Up to 42 months
  DOR defined as time from study entry to change in response from CR or PR to Stable Disease (SD) or Progressive Disease (SD) (as assessed by RECIST v1.1).
To assess the safety and tolerability of the combination of cabozantinib and one-week-on one-week-off temozolomide | Up to 42 months
  Safety and tolerability as assessed by adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0.
  After five patients, it will be perform a detailed safety report based on CTCAE v.5.0
To assess the predictive role of MGMT Methylation Status on response to the combination of cabozantinib and one-week-on one-week-off temozolomide | Up to 42 months
  MGMT Methylation Status will be assessed and any correlation with the efficacy endpoints will be evaluated.
To assess the activity of the combination of cabozantinib and one-week-on one-week-off temozolomide at 1 year from the start of the treatment | 1 year overall survival OS
  1 year overall survival OS

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Institute of Naples, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: No